CLINICAL TRIAL: NCT01415817
Title: The Effect of an Intensive Endoscopic Quality Improvement Program (EQUIP) on Improved Detection and Classification of Non-polypoid (Flat and Depressed) and Polypoid Colorectal Adenomas. ("EQUIP" Study)
Brief Title: Endoscopic Quality Improvement Program
Acronym: EQUIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Michael B. Wallace, Mayo Clinic Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10-000433
Record Dates: First submitted 2011-08-08; First posted 2011-08-12 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Adenomatous Polyps; Colorectal Polyps
Keywords: Quality Improvement; Adenoma Detection Rate; Polyp detection rate; Colonoscopy; Training; Colorectal cancer screening
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline Data collection (No Intervention)
- Randomization and Training Arm (Experimental)
  Interventions: Other: Training session

INTERVENTIONS:
Other: Training session — Series of two training sessions after the first phase of study followed by monthly feedback.
  Arms: Randomization and Training Arm

SUMMARY:
Effective colorectal cancer (CRC) screening relies on early identification and removal of both polypoid and non-polypoid lesions with neoplastic potential. The investigators hypothesize that an intensive training program designed to enhance both recognition and classification of lesions with neoplastic potential, will result in an increase in non-polypoid adenoma detection in addition to and independent of an increase in overall adenoma detection rates.

DETAILED DESCRIPTION:
Our Endoscopic Quality Improvement Program (EQUIP) was a prospective educational intervention with our staff endoscopist as our study population. The investigators measured adenoma detection rates for a baseline period then randomly assigned half of the endoscopists to undergo EQUIP training. The investigators then examined baseline and post-training study adenoma detection rates (ADR's) for all endoscopist (trained and un-trained) to evaluate the impact of training.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopies performed at Mayo clinic ambulatory surgical center

Exclusion Criteria:

* Procedures for the indication of acute GI hemorrhage
* Active colitis
* Hereditary polyposis syndrome
* Inflammatory bowel disease
* Incomplete procedures
* Procedures with surgically altered anatomy (i.e. prior colectomy)
* Poor bowel preparation (Boston Bowel preparation score <5) were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measurement of overall adenoma detection rate | 1 year
  Primary outcome measures will include overall and per patient adenoma detection rate for polypoid and non polypoid neoplastic lesions.

SECONDARY OUTCOMES:
Measurement of total polypectomy rate | 1 Year
  Secondary outcomes will include total polypectomy rate (hyperplastic vs. adenoma),
Measurement of colonoscopy time | 1 Year
  Total colonoscopy time and endoscopist acceptance. Variables such as patient demographics and prep quality will be adjusted for.
Endoscopist Acceptance | 1 Year
  Ensdoscopist acceptance rate will be measured. Variables such as patient demographics and prep quality will be adjusted for.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Wallace, MD,MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States